CLINICAL TRIAL: NCT03725215
Title: Influence of Multiple Ratio Split-belt Treadmill on Gait Asymmetry and Motor Learning in PD Patients With Freezing of Gait
Brief Title: Motor Adaptation to Split-Belt Treadmill in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: University of Kiel (Other)
Responsible Party: Principal Investigator, Alice Nieuwboer, Senior Professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S60876
Record Dates: First submitted 2018-07-12; First posted 2018-10-30 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Parkinson Disease; Freezing of Gait
Keywords: Split-Belt Treadmill; Training
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Participants will randomly be assigned to 1 of 4 different split-belt treadmill paradigms. Assessments will be performed pre and post training on day 1 and once again on day 2.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Split-Belt Treadmill Training 1:2 (Experimental): Split-Belt Training with a steady ratio of 1:2.
  Interventions: Behavioral: Split-Belt Treadmill Training
- Split-Belt Treadmill Training 3:4 (Experimental): Split-Belt Training with a steady ratio of 3:4.
  Interventions: Behavioral: Split-Belt Treadmill Training
- Split-Belt Treadmill Training Changing (Experimental): Split-Belt Training with changing ratios between 3:4 to 1:2.
  Interventions: Behavioral: Split-Belt Treadmill Training
- Split-Belt Treadmill Training Tied-Belt (Active Comparator): Split-Belt Training with tied belts.
  Interventions: Behavioral: Split-Belt Treadmill Training

INTERVENTIONS:
Behavioral: Split-Belt Treadmill Training — One session of 6 x 5 min with 1 min intervals.

SUMMARY:
Freezing of Gait (FOG) is a disabling symptom common in advanced Parkinson's Disease. FOG is an independent contributor to fall risk and is only partially relieved by medication. Parkinson's patients with FOG are known to have more difficulty with gait adaptation in their day to day environment. Further, asymmetry of gait has been implicated in FOG as these episodes are often elicited during asymmetric tasks such as turning. This study will examine the effect of a single session of split-belt treadmill walking on gait adaptation, gait symmetry and FOG as well as 24 hour retention of these effects.

DETAILED DESCRIPTION:
In this proposal, the investigators will investigate whether adapting gait to modulations imposed by a split-belt treadmill, improves walking ability and reduces FOG. The investigators will test the hypothesis that motor adaptation deficits underlie FOG and that these problems are modifiable with training. To address these suppositions, the investigators propose a multi-centric study conducted in two research labs with expertise in split-belt gait analysis and FOG: University of Leuven (KUL) and Christian-Albrechts-University Kiel (CAUK). As freezers have been shown to have more difficulty with consolidation of motor learning, the investigators aim in study I (pilot phase) to first understand which split-belt parameters are optimal for training gait flexibility and lead to consolidated gains in daily walking. For this study, the investigators will recruit 60 freezers and 60 healthy controls, pooled across centers, and manipulate different split-belt conditions in one learning and retention session.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's Disease as per the UK Parkinson's Disease Society Brain Bank Criteria
* Classification as a Freezer with the New Freezing of Gait Questionnaire (score > 0)
* Ability to walk at least 5 min. without any aid
* Stable anti-parkinsonian medication at least 1 month prior to participation

Exclusion Criteria:

* Neurologic diseases other than PD
* Orthopedic injuries that could influence gait and balance
* Participation in treadmill training more than once a week
* Cognitive impairment (MMSE<24) or inability to follow test instructions
* Self-reported DBS-related postural or gait disturbances
* Cardiovascular risk factors
* Peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Adaptation to Split/Tied Belt | 24 hours after training
  Measured with 3D motion analysis system during treadmill walking. Patients will walk for 1.5 minutes on the treadmill that will switch from tied-to-split state and back to tied state.
Gait Asymmetry | 24 hours after training
  Measured with 3D motion analysis system during straight line overground walking
Freezing Ratio | 24 hours after training
  Measured with APDM sensors during 360 degree turns

SECONDARY OUTCOMES:
Medio-lateral Anticipatory Postural Adjustments | 24 hours after training
  Measured with APDM sensors at gait initiation
Gait Speed during dual task walking | 24 hours after training
  Measured with 3D motion analysis system during overground walking with an auditory Stroop task

CONTACTS AND LOCATIONS:
Overall Officials: Alice Nieuwboer, PhD, Principal Investigator — KU Leuven; Christian Schlenstedt, PhD, Principal Investigator — CAU Kiel
Locations (2):
- Faculty of Movement and Rehabilitation Sciences (FaBeR), Leuven, Belgium
- University Hospital Schleswig-Holstein, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seuthe J, D'Cruz N, Ginis P, Becktepe JS, Weisser B, Nieuwboer A, Schlenstedt C. The Effect of One Session Split-Belt Treadmill Training on Gait Adaptation in People With Parkinson's Disease and Freezing of Gait. Neurorehabil Neural Repair. 2020 Oct;34(10):954-963. doi: 10.1177/1545968320953144. Epub 2020 Sep 17. PMID 32940131

DOCUMENTS (1):
  • Study Protocol (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT03725215/Prot_000.pdf